CLINICAL TRIAL: NCT04473482
Title: Michigan Alcohol Improvement Network- Alcohol Reduction and Treatment Trial
Acronym: MAIN-ART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Jessica Mellinger, Assistant Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00174946; 5K23AA026333-02 (NIH)
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Results first posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Alcohol-Related Disorders; Liver Diseases
MeSH Terms: conditions — Alcohol-Related Disorders; Liver Diseases | interventions — Ethanol

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MAIN-ART Behavior Tool (Experimental): The Michigan Alcohol Improvement Network- Alcohol Reduction and Treatment Tool (MAIN-ART) behavioral intervention is an online web application with two modules: misconception correction and tailored, preference-sensitive alcohol use disorder (AUD) treatment matching.
  Interventions: Behavioral: Michigan Alcohol Improvement Network-Alcohol Reduction and Treatment tool
- Routine care (No Intervention): Patients randomized to usual care will receive a pamphlet for alcohol treatment referral to the University of Michigan Addiction Treatment Services, but will receive no further education from the research team.

INTERVENTIONS:
Behavioral: Michigan Alcohol Improvement Network-Alcohol Reduction and Treatment tool — The intervention corrects misconceptions about alcohol use, liver disease, and alcohol treatment and matches patients to their top three choices of treatment while providing them with brief explanations of each treatment option.
  Arms: MAIN-ART Behavior Tool

SUMMARY:
The purpose of the study is to determine if providing participants with alcohol-related liver disease with tailored alcohol use treatment options is feasible and acceptable in order to increase their engagement with treatment and reduce alcohol use. This is an important area to study to help create ways to increase participants' knowledge about different treatment options as well as increase likelihood of seeking and participating in alcohol use disorder treatments.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled at University of Michigan general hepatology clinics or inpatient wards
* Documented diagnosis of alcohol-associated cirrhosis or alcoholic hepatitis or alcohol-related liver disease of any stage
* Drinking of any amount of alcohol within the 6 months prior to recruitment
* No alcohol use treatment within the past 1 month
* Access to a phone for purposes of follow-up

Exclusion Criteria:

* Active alcohol use treatment
* Undergoing active evaluation for liver transplantation, is listed for liver transplant, or is post-transplantation.
* Is enrolled in the multidisciplinary alcohol-related liver disease clinic at Michigan Medicine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Mellinger, MD, MSc, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mellinger JL, Medley S, Kidwell KM, Asefah H, Winder GS, Fernandez AC, Lok ASF, Blow F. Improving alcohol treatment engagement using integrated behavioral interventions in alcohol-associated liver disease: A randomized pilot trial. Hepatol Commun. 2023 Sep 15;7(10):e0181. doi: 10.1097/HC9.0000000000000181. eCollection 2023 Oct 1. PMID 37708435

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MAIN-ART Behavior Tool | Routine Care
Started | 30 | 30
3-month Post Intervention Phone Call | 22 | 27
6-month Post Intervention Phone Call | 19 | 19
Completed | 19 | 19
Not Completed | 11 | 11
Not completed — Death | 0 | 3
Not completed — Lost to Follow-up | 9 | 7
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MAIN-ART Behavior Tool | Routine Care | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (11.3) | 50.0 (13.4) | 48.4 (12.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 15 | 15 | 30
  Gender: Male | 15 | 15 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 24 | 27 | 51
  Black | 3 | 1 | 4
  Native American | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Unknown/Declined to Answer | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 30 | 60
Alcohol-Related Liver Disease (ALD) Severity [Count of Participants; unit: Participants]
  Alcohol related cirrhosis or acute alcohol related hepatitis or both | 23 | 20 | 43
  Alcohol-related Steatosis | 7 | 10 | 17
Cirrhosis Diagnosis [Count of Participants; unit: Participants]
  Compensated Cirrhosis | 3 | 4 | 7
  Decompensated Cirrhosis | 17 | 13 | 30
  Alcohol-Related Liver Disease (ALD), No Cirrhosis | 10 | 13 | 23
Self-reported last drink [Mean (Standard Deviation); unit: Days] | 60 (11.2) | 61 (12.4) | 60.5 (11.7)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of MAIN-ART Tool as Measured by Recruitment Rates
Description: Feasibility of administration of the MAIN-ART tool will be determined by recruitment rates and retention rates (as measured at 6 months after recruitment). Study recruitment started on 23 September, 2020 and concluded on 10 January 2022. The results reflect the number and percent of those patients who were approached, were determined to be eligible, and were consented.
Time Frame: Up to 6 months
Population: This population is prior to consent and includes the patients who were ultimately excluded due to not meeting study criteria, cancellation, not showing up to appointments, being unreachable via phone, or for declining participation in the study.
Measure: Count of Participants; unit: Participants
Groups:
- Clinical Population: Patients in hepatology and the University of Michigan Hospital's inpatient ward who were approached about possible participation in this study.
Arm/Group | Clinical Population
Number analyzed (Participants) | 276
Participants | 60

2. Primary Outcome: Feasibility of MAIN-ART Tool as Measured by Retention Rates
Description: Feasibility of administration of the MAIN-ART tool will be determined by recruitment rates and retention rates (as measured at 6 months after recruitment). Retention rate is shown by the number of participants who continued in the study for 6 months, and the percentage that it represents compared to those who began it but did not follow through to the end of the study (6 months).
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | MAIN-ART Behavior Tool | Routine Care
Number analyzed (Participants) | 30 | 30
Participants | 19 | 19

3. Primary Outcome: Acceptability of the MAIN-ART Tool as Measured by Post-intervention Surveys
Description: On the day the participants engage with the MAIN-ART tool, acceptability will be determined by patient-level surveys. The System usability Survey (SUS) consists of 10 questions ranging from 1 (strongly disagree) to 5 (strongly agree). A scoring algorithm which produces a range from 0 to 100 was used. Current literature suggests that a score above 68 for mean SUS is considered "above average." By "intervention," this measure means interaction with the MAIN-ART tool, which occurs only at the participant's initial visit.
Time Frame: Up to 1 hour
Population: Only subjects randomized to the intervention MAIN-ART behavioral tool were assessed in the intervention group. Because this intervention was given at the initial visit, all participants who were randomized to the MAIN-ART tool arm are available for analysis.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | MAIN-ART Behavior Tool
Number analyzed (Participants) | 30
score on a scale | 70 [47.5 to 95]

4. Secondary Outcome: Alcohol Use Frequency as Measured by the Alcohol Timeline Follow-back (TLFB) Interview
Description: Alcohol use will be defined according to World Health Organization (WHO) risk drinking level. WHO drinking risk levels were derived from patient reports of the number of standard drinks (defined as 0.6 ounces of absolute alcohol) consumed, which were converted to grams of pure alcohol (0.6 ounces = 14 grams). Ranging from abstinence (0 grams) to very high risk (101+ males / 61+ females grams).
Time Frame: Baseline and 6 months
Population: Baseline measure data includes all participants whose data was collected at baseline. The participants at 6 months includes only those who completed the study.
Measure: Mean (Standard Deviation); unit: Grams per day
Arm/Group | MAIN-ART Behavior Tool | Routine Care
Number analyzed (Participants) | 30 | 30
Grams per day
  Baseline | 87 (192) | 72 (191)
  6 months: number analyzed (Participants) | 19 | 19
  6 months | 13 (33) | 29 (75)
Statistical Analysis 1: Comparison: MAIN-ART Behavior Tool vs Routine Care; Test type: Superiority — Generalized estimating equations with robust sandwich estimators used with Wald 95% confidence intervals and conversion to odds ratios; Odds Ratio (OR) = 2.25 — Generalized estimating equations with robust sandwich estimators used with Wald 95% confidence intervals and conversion to odds ratios; Generalized estimating equations with robust sandwich estimators used with Wald 95% confidence intervals

5. Secondary Outcome: Alcohol Treatment Engagement as Measured by Number of Participants Who Engaged in Any Alcohol Cessation or Reduction Visit as Measured by Self-report.
Description: Alcohol treatment engagement will be defined as at least one visit with formal, external assistance in alcohol cessation or reduction including inpatient rehabilitation services, out patient alcohol cessation programs, engagement in therapy of any kind tailored for alcohol cessation, and engagement in any group therapy or support groups for alcohol cessation including alcoholics anonymous, 12 step facilitation and etc.
Time Frame: Up to 6 months
Population: All participants involved in the initial use of the MAIN-ART tool or who received routine care are analyzed to evaluate what percent engaged with alcohol treatment by the end of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | MAIN-ART Behavior Tool | Routine Care
Number analyzed (Participants) | 30 | 30
Participants | 8 | 4
Statistical Analysis 1: Comparison: MAIN-ART Behavior Tool vs Routine Care; Test type: Superiority; Odds Ratio (OR) = 2.31 — GEEs with robust sandwich estimators and Wald 95% CIs with conversion to Odds Ratios

ADVERSE EVENTS:
Time Frame: Up to 6 months.
Arm/Group | MAIN-ART Behavior Tool | Routine Care
All-Cause Mortality (participants affected / at risk) | 0/30 | 3/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-18): https://cdn.clinicaltrials.gov/large-docs/82/NCT04473482/Prot_SAP_001.pdf
  • Informed Consent Form (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/82/NCT04473482/ICF_000.pdf